CLINICAL TRIAL: NCT07147712
Title: Interventions to Promote Well-being and Social Relationships Among University Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1232-b
Record Dates: First submitted 2025-07-18; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-05

CONDITIONS: Loneliness; Psychological Well Being; Social Relationship
Keywords: university students; well being; social relationships; socialization
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study will use a randomized controlled design to test the impact of a brief psychological group intervention on university students' psychological well-being and social connectedness. Participants will be randomly assigned to either the intervention group (immediate participation in the 6-session program) or the control group (waitlist, intervention after follow-up).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - Psychological Group Intervention (Experimental): Intervention Group (receives the program immediately)
  Interventions: Behavioral: Psychological Group Intervention
- Control group - waitlist (No Intervention): Participants in the waitlist control group will not take part in the intervention during the initial phase of the study. They will complete all assessments at the same time points as the experimental group (pre, post, and follow-up) and will be offered the same 6-session intervention after the follow-up data collection is complete.

INTERVENTIONS:
Behavioral: Psychological Group Intervention — 6-session psychological group intervention, delivered once per week over six weeks. The intervention is designed to promote well-being and improve the quality of social relationships. It includes psychoeducational content, experiential exercises, and guided group discussions focused on emotional expression, social connection, and mutual support. A follow-up session will be offered after 4 weeks. Sessions will be led by trained psychologists and conducted in a university setting.
  Arms: Experimental - Psychological Group Intervention

SUMMARY:
This study evaluates the impact of a psychological group intervention aimed at promoting well-being and social connectedness among university students. The intervention is part of the UNIST-HEALTH (PRO-BEN) initiative and targets students enrolled at the University of Padua. Participants will be randomly assigned to either an intervention group or a waitlist control group. The intervention consists of six weekly group sessions focused on psychoeducation and experiential activities designed to enhance the quality of social relationships, reduce loneliness, and improve psychological well-being. Assessments will be conducted at baseline, post-intervention, and at a four-week follow-up.

DETAILED DESCRIPTION:
University students are a population at heightened risk for psychological distress, with increasing levels of loneliness, anxiety, and depression reported globally. The university period represents a developmental transition characterized by academic, social, and emotional challenges.

Extensive research has shown that strong social relationships are critical to psychological well-being. High levels of social connectedness are associated with lower rates of anxiety and depression, and promote greater life satisfaction, emotional resilience, and academic adjustment. In contrast, loneliness and perceived social isolation are predictors of psychological distress and negative health outcomes.

To address these issues, the aim of this study is to evaluate the impact of a brief psychological group intervention designed to promote well-being and enhance the quality of social relationships among university students. The intervention is developed within the framework of the UNIST-HEALTH (PRO-BEN) project.

Assessment Phase The study begins with an initial screening phase. Participants are invited to attend a brief individual interview with a trained psychologist to assess their psychological health status, motivation to participate, and expectations regarding the intervention.

Following the interview, participants complete a baseline questionnaire collecting demographic information (e.g. age, gender, course of study, country of origin, type of housing - 10 questions) and measures from self-report instruments, including:

* Questions regarding health status and social life (e.g. social and sports activities practiced) - 11 questions.
* UCLA Loneliness Scale - 3-item version: 3 items to measure subjective feelings of loneliness and social isolation.
* Psychological Well-Being Scale: 18 items to measure psychological well-being.
* General Anxiety Disorder-7: 7 questions about the perception of anxious symptoms in the last two weeks.
* Patient Health Questionnaire-9: 9 questions about the frequency with which, in the last two weeks, different problems attributable to depressive symptoms have been faced.
* Work and Social Adjustment Scale: 5 questions about functioning in social and work life.
* Multidimensional Scale of Perceived Social Support: 12 questions to measure perceived support, in particular from friends, family and partners.
* Sense of community: brief scale developed ad hoc to evaluate perception of belongingness to different groups

Participants complete the same set of questionnaires at three time points:

* Baseline (pre-intervention)
* Post-intervention (after 6 weeks)
* Follow-up (4 weeks after the final session) Intervention Phase Eligible participants are randomly assigned to either the intervention group or the control group (waitlist). The intervention group will immediately take part in a 6-session group-based program (one session per week, for six consecutive weeks), while the control group will receive the same intervention only after the follow-up period has been completed. Sessions will include psychoeducational modules, experiential exercises, and guided group discussions.

The study aims:

* to assess the feasibility and acceptability of a 6-weeks intervention to promote psychological and general well-being on university students
* to assess the impact of the intervention compared to a control group who did not receive it

ELIGIBILITY:
Inclusion Criteria:

* University students regularly enrolled at the University of Padua
* Aged 18 years or older
* Able to understand and complete the questionnaires in Italian or English
* Residing in Padova or its province during the study period
* Providing informed consent for participation

Exclusion Criteria:

* Presence of severe psychological conditions requiring immediate or specialized clinical care, as identified during the initial screening interview
* Inability or unavailability to attend group sessions for the full 6-week duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Between group differences (experimental vs control group) in wellbeing levels | baseline, 6-weeks, 4-weeks follow-up
  Psychological Well-Being Scale (PWS; min=18, max=108; higher scores indicate greater wellbeing)
Between group differences (experimental vs control group) in loneliness levels | baseline, 6-weeks, 4-weeks follow-up
  UCLA Loneliness Scale - 3-item version (min=3, max=9; higher scores indicate higher levels of loneliness)
Adherence to the intervention | 6-weeks, 4-weeks follow-up
  Participants' attendance rates to the sessions
Acceptability of the intervention | 6-weeks
  Participants' rates to the satisfaction questionnaire, developed ad hoc for the present study (min=8, max= 56; higher scores indicate higher satisfaction)

SECONDARY OUTCOMES:
Between group differences (experimental vs control group) in symptoms of anxiety | baseline, 6-weeks, 4-weeks follow-up
  General Anxiety Disorder-7 (GAD-7). Higher scores indicate greater anxiety severity (min=0, max=21)
Between group differences (experimental vs control group) in symptoms of depression | baseline, 6-weeks, 4-weeks follow-up
  Patient Health Questionnaire-9 (PHQ-9). A higher score means more severe symptoms (min=0, max=27)

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Padova, Padua, Padova, Italy

IPD SHARING:
Plan to Share IPD: No
A plan will be established by the research team for data sharing following publication of the first manuscript

REFERENCES:
- [Background] Cipolletta S, Tedoldi I, Tomaino SCM. A blended group intervention to promote social connectedness and wellbeing among international university students: an exploratory study. Front Psychol. 2024 Nov 27;15:1497544. doi: 10.3389/fpsyg.2024.1497544. eCollection 2024. PMID 39664633